CLINICAL TRIAL: NCT03136848
Title: A Single Centre Study of the Feasibility and Safety of Using Normothermic ex Vivo Machine Perfusion to Store Human Kidneys for Transplantation.
Brief Title: The Feasibility and Safety of Normothermic ex Vivo Kidney Perfusion
Acronym: NEVKP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-9907-A
Record Dates: First submitted 2017-03-08; First posted 2017-05-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-03

CONDITIONS: Kidney Transplantation
Keywords: perfusion

STUDY DESIGN:
Intervention Model Description: A pilot study of procedural feasibility involving both device and drug (organ perfusate solution).
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normothermic perfusion (Experimental): Kidneys retrieved from deceased donors will undergo the study intervention consisting of 4-10 hours of Normothermic ex-vivo perfusion using a blood-based solution, prior to implantation in the transplant recipient
  Interventions: Drug: Normothermic ex-vivo kidney perfusion Solution -Toronto

INTERVENTIONS:
Drug: Normothermic ex-vivo kidney perfusion Solution -Toronto — The perfusion "device" will circulate warmed, oxygenated blood-based perfusate ("Normothermic ex-vivo kidney perfusion solution-Toronto") through the kidney.

SUMMARY:
Kidney transplantation is the treatment of choice for end-stage kidney failure, but access to transplantation is limited by a severe shortage of donor organs. Although the use of kidneys from higher risk deceased donors has increased the availability of organs, these grafts are associated with a greater risk of delayed function, inferior performance, and shorter survival than standard criteria donor kidneys. The current standard of care for kidney graft preservation prior to transplantation is static cold storage. Preliminary results from large animal kidney transplantation studies and a human clinical trial suggest that normothermic machine perfusion of kidneys prior to transplantation may ameliorate the injury sustained by kidney grafts during cold static preservation, allow assessment of organ viability prior to transplantation, and reduce the risk of delayed graft function or non-function. Such a strategy may not only improve the performance of kidneys that are currently considered acceptable for transplantation, but may also facilitate the assessment and utilization of kidneys that are currently not considered for transplantation. This study will examine the feasibility and safety of normothermic ex vivo perfusion of human kidneys prior to transplantation. The study will evaluate kidney function after transplantation using standard clinical parameters. Study participants will be followed for 3 months following transplantation and their outcomes recorded. Feasibility will be measured using the ratio of actual:eligible kidney grafts preserved by normothermic ex vivo perfusion and will also take into account logistical issues with respect to implementation and ease of use of the ex vivo perfusion device. Safety will be assessed by rates of device failure resulting in organ discard, primary graft non-function, delayed graft function, graft failure, and recipient mortality.

DETAILED DESCRIPTION:
Kidney transplantation is the treatment of choice for suitable patients with end-stage renal disease as it results in lower morbidity and mortality rates when compared to dialysis. Unfortunately, the number of patients referred for transplantation has grown more quickly than the number of suitable grafts from deceased donors.

The use of higher risk organs has expanded the donor pool but at a great cost due to the higher probability that higher risk kidneys will never function (primary non-function, PNF), or will have delayed graft function (DGF). The current standard of care for kidney graft preservation prior to transplantation is static cold storage but higher-risk deceased donor kidneys are particularly vulnerable to the effects of cold storage. Preliminary results from large animal kidney transplantation studies and a human clinical trial suggest that normothermic machine perfusion of kidneys prior to transplantation may ameliorate the injury sustained by kidney grafts during cold static preservation, allow assessment of organ viability prior to transplantation, and reduce the risk of delayed graft function or non-function. Such a strategy may not only improve the performance of kidneys that are currently considered acceptable for transplantation, but may also facilitate the assessment and utilization of kidneys that are currently not considered for transplantation.

This study will examine the feasibility and safety of normothermic ex vivo perfusion of human kidneys prior to transplantation. Kidneys will be retrieved in the standard fashion and stored cold during transit. Upon arrival at the study transplant centre, kidneys will begin perfusion with a normothermic near-physiologic, blood-based solution. Perfusion will last 1-10 hours.

The study will evaluate kidney function after transplantation using standard clinical parameters. Study participants (n=25) will be followed for 3 months following transplantation and their outcomes recorded. Feasibility will be measured using the ratio of actual:eligible kidney grafts preserved by normothermic ex vivo perfusion and will also take into account logistical issues with respect to implementation and ease of use of the ex vivo perfusion device. Safety will be assessed by rates of device failure resulting in organ discard, primary graft non-function, delayed graft function, graft failure, and recipient mortality.

ELIGIBILITY:
Inclusion Criteria (Organ):

* Single kidneys from DBD (donation after brain death) and DCD (donation after cardiac death) donors
* Kidney is subjected to a maximum of 12 hours of cold storage prior to beginning of NEVKP (normothermic ex vivo kidney perfusion)
* Kidney meets parameters that are acceptable for transplantation according to the study transplant centre's current clinical practices.

Exclusion Criteria (Organ):

* Kidneys from living donors
* Kidneys that would be declined for transplantation under the study centre's current clinical practice
* Kidneys with multiple arteries.
* Kidney grafts from donors positive for Hepatitis B surface antigen or Hepatitis C viremia.

Inclusion Criteria (Participants):

• Adult male and female patients (18 years or more), active on the waiting list for kidney transplantation; able to give informed consent.

Exclusion Criteria (Participants):

* Patients with focal segmental glomerulosclerosis (FSGS)
* Patients with a diagnosis of atypical hemolytic uremic syndrome, membranoproliferative glomerulonephritis, or thrombotic microangiopathy Patients with a calculated Panel Reactive Antibody (cPRA) greater than 95%
* Patients with known allergies to any of the perfusion solution components
* Patients undergoing retransplantation
* Recipients with pre-existing vascular disease posing technical challenges for transplantation
* Recipients with any clinically-relevant positive DSA (donor-specific antibody) identified
* Transplantation of more than one organ (e.g. liver/pancreas and kidney)
* Refusal of informed consent
* Recipients receiving double kidney grafts (i.e. both kidneys from one donor being transplanted into a single recipient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
the ratio of actual / eligible kidney grafts subjected to study intervention. | assessed 3 months after enrollment of final participant, or up to 48 months, whichever is earlier
  planned versus actual kidney perfusions to assess study feasibility
The rate of kidney discard or graft failure attributable to the study intervention | from date of first actual intervention to date last participant completes the study followup period of 3 months post-intervention
  organ discard or graft failure directly attributable to the use of normothermic perfusion

SECONDARY OUTCOMES:
duration of post-transplant dialysis | 3 months post-kidney transplantation
rate of primary graft non-function compared to historical, case-matched controls | 3 months post-kidney transplantation
Degree of Ischemia-reperfusion injury as assessed by post-reperfusion kidney biopsies | assessed 3 months after enrollment of final participant
  Pre--implantation kidney biopsies will be graded according to standard histological criteria and assess for degree of ischemia-reperfusion injury
Rate of delayed graft function | 3 months post-kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Markus Selzner, MD, Principal Investigator — Surgeon, MOT, UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazilescu LI, Urbanellis P, Kim SJ, Goto T, Noguchi Y, Konvalinka A, Reichman TW, Sayed BA, Mucsi I, Lee JY, Robinson LA, Ghanekar A, Selzner M. Normothermic Ex Vivo Kidney Perfusion for Human Kidney Transplantation: First North American Results. Transplantation. 2022 Sep 1;106(9):1852-1859. doi: 10.1097/TP.0000000000004098. Epub 2022 Mar 1. PMID 35238854